CLINICAL TRIAL: NCT03769662
Title: XT-150-1-0201 Extension: Evaluation of Safety, Tolerability, and Efficacy of XT-150 for the Treatment of Osteoarthritic Pain
Brief Title: Follow on Extension of XT-150-1-0201
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xalud Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XT-150-1-0203
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-12

CONDITIONS: Osteoarthritis, Knee
Keywords: Cytokines; Anti-inflammatory; Pain; Inflammation
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Inflammation

STUDY DESIGN:
Intervention Model Description: Open-label, single dose study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- High dose from study XT-150-1-0201 (Experimental): Open label administration of the highest dose in the earlier study, in which all doses were well tolerated
  Interventions: Biological: XT-150

INTERVENTIONS:
Biological: XT-150 — IL-10 transgene DNA plasmid injected into the knee synovial capsule

SUMMARY:
XT-150 safety and efficacy in severe osteoarthritic pain.

DETAILED DESCRIPTION:
XT-150-1-0201 Extension: Evaluation of Safety, Tolerability, and Efficacy of XT-150 for the Treatment of Osteoarthritic Pain.

Participants in this study will have been enrolled in the 0201 study and qualify for an intra-articular injection of XT-150 into the osteoarthritic knee.

The study will assess XT-150 safety, tolerability, and efficacy in participants who received placebo in the 0201 study, or have a second qualifying knee, or a second injection into the same knee that was treated in 0201.

ELIGIBILITY:
Inclusion Criteria:

1. Qualified and participated in clinical study XT-150-1-0201.

   1. Participant was assigned to placebo, or
   2. Participant elects to have XT-150 administered to the XT-150-untreated knee that qualified under XT-150-1-0201 criteria, or
   3. Participant had inadequate pain relief and elects to receive a second injection to the same knee treated on clinical study XT-150-1-0201
2. Sufficiently severe OA of knee to require/have recommended knee replacement surgery or be unsuitable for knee replacement surgery based on co-morbidities or orthopedic considerations; be free of local or intra-articular infection.
3. Symptomatic disease because of osteoarthritis, defined as a Verbal Numerical Rating Scale (VNRS) scores of a worst pain of at least 7 at any time during the preceding week (based on scale of 0 to 10, with 10 representing "pain as bad as you can imagine").
4. Stable analgesic regimen during the 4 weeks prior to enrollment.
5. Inadequate pain relief (minimum ≥ 5 mean on Brief Pain Inventory-Severity Scale) lasting more than 3 months.
6. In the judgment of the Investigator, acceptable general medical condition
7. Life expectancy >6 months
8. Male participants who are heterosexually active and not surgically sterile must agree to use effective contraception, including abstinence, for the duration of the study and for 3 months after the study is completed.
9. Have suitable knee joint anatomy for intra-articular injection
10. Willing and able to return for the follow-up (FU) visits
11. Able to reliably provide pain assessment
12. Able to read and understand study instructions, and willing and able to comply with all study procedures

Exclusion Criteria:

1. Hypersensitivity, allergy, or significant reaction to any ingredient of the study drug, including double-stranded DNA, mannose, and sucrose
2. Scheduled knee replacement within 4 months; participant agrees not to schedule a knee replacement appointment within 4 months of study treatment
3. History of rheumatoid arthritis of the knee or gout.
4. High peri-operative risks which in the judgment of the investigator preclude a safe knee injection procedure (e.g., poorly controlled diabetes, cardiac inadequacy such as NYHA class > II, G4 glomerular filtration rate [eGFR < 30 mL/min by Cockcroft-Gault])
5. Current treatment with immunosuppressive (systemic corticosteroid therapy [equivalent to >10mg/day prednisone] or other strong immunosuppressant)
6. History of immunosuppressive therapy; high-potency systemic steroids in the last 3 months.
7. Currently receiving systemic chemotherapy or radiation therapy for malignancy
8. Clinically significant hepatic disease as indicated by clinical laboratory results ≥3 times the upper limit of normal for any liver function test (e.g., aspartate aminotransferase, alanine aminotransferase, lactate dehydrogenase)
9. Severe anemia (Grade 3; hemoglobin <8.0 g/dL, <4.9 mmol/L, <80 g/L; transfusion indicated), uncontrolled coagulopathy (Grade 1, prolonged activated partial prothrombin time (aPTT) > upper limit of normal (ULN) to 1.5xULN), or bleeding diathesis, Grade 1 white cell counts (lymphocytes <LLN - 800/mm3; <LLN - 0.8 x 109 /L, neutrophils <LLN - 1500/mm3; <LLN - 1.5 x 109 /L)
10. Significant neuropsychiatric conditions; dementia, major depression, or altered mental state that in the opinion of the Investigator will interfere with study participation
11. Current treatment with systemic antibiotics or antivirals (EXCEPTION: topical treatments)
12. Current treatment with anticoagulants, other than low-dose aspirin.
13. Known or suspected history of active alcohol or intravenous/oral drug abuse within 1 year before the screening visit
14. Women of child-bearing potential
15. Use of any investigational drug, other than XT-150, or device within 1 month before enrollment or current participation in a trial that included intervention with a drug or device; or currently participating in an investigational drug or device study.
16. Any condition that, in the opinion of the Principal Investigator, could compromise the safety of the participant, the participant's ability to communicate with the study staff, or the quality of the data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 6 months
  Clinical Pathology, adverse events

SECONDARY OUTCOMES:
Verbal Numeric Rating Score | 6 months
  Pain scale from 1 to 10, 10 being worst possible
KOOS | 6 months
  Osteoarthritis pain, symptoms, impact on daily living, and quality of life. Subset scores are calculated such that 100% is normal function
Brief Pain Inventory | 6 months
  Pain and interference on daily living functions. Scales ranges from 0 to 10, with 10 being the worst
Clinical Global Improvement | 6 months
  0 - 7 Scale, 4 and below indicate no change or improvement. Over 4 indicates degrees of worsening

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rickman, MD, Principal Investigator — University of Adelaide
Locations (1):
- CMAX Clinical Research Pty Ltd in collaboration with University of Adelaide, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No